CLINICAL TRIAL: NCT00451100
Title: Comparison of Rocuronium and Org25969 With Cisatracurium and Neostigmine When Neuromuscular Block is Reversed at Reappearance of T2
Brief Title: Comparison of Rocuronium and Org 25969 With Cisatracurium and Neostigmine (19.4.310)(P05931)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05931; Crystal Trial; 19.4.310
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex (Experimental): 2.0 mg/kg Org 25969 (sugammadex)
  Interventions: Drug: Sugammadex
- Neostigmine (Active Comparator): 50 ug/kg neostigmine
  Interventions: Drug: neostigmine

INTERVENTIONS:
Drug: Sugammadex — Subjects received a bolus dose of 0.6 mg/kg rocuronium. After the last dose of rocuronium, at reappearance of T2, a dose of 2.0 mg/kg Org 25969 was to be administered
  Other Names: Org 25969
  Arms: Sugammadex
Drug: neostigmine — Subjects received a bolus dose of 0.15 mg/kg cisatracurium. After the last dose of cisatracurium, at reappearance of T2, a dose of 50 ug/kg neostigmine was to be administered. In accordance to the labeling of neostigmine, a maximum of 5 mg neostigmine was to be administered
  Other Names: premix neostigmine/glycopyrrolate
  Arms: Neostigmine

SUMMARY:
The purpose of this study was to demonstrate in adult patients a faster recovery from a neuromuscular block with 2.0 mg/kg Org 25969 (sugammadex) after rocuronium as compared to 50 ug/kg neostigmine after cisatracurium when administered at reappearance of T2

ELIGIBILITY:
Inclusion Criteria:

* Subjects of ASA 1 - 4;
* Subjects above or equal to the age of 18;
* Scheduled for surgical procedures with a general anesthesia requiring neuromuscular relaxation with the use of rocuronium or cisatracurium;
* Scheduled for surgical procedures in supine position;
* Given written informed consent.

Exclusion Criteria:

* Subjects in whom a difficult intubation because of anatomical malformations was expected;
* Subjects known or suspected to have neuromuscular disorders impairing neuromuscular block (NMB) and/or significant renal dysfunction;
* Subjects known or suspected to have a (family) history of malignant hyperthermia;
* Subjects known or suspected to have an allergy to narcotics, muscle relaxants or other medication used during general anesthesia;
* Subjects receiving medication in a dose and/or at a time point known to interfere with neuromuscular blocking agents such as antibiotics, anticonvulsants and Mg2+;
* Subjects in whom the use of neostigmine and/or glycopyrrolate may be contraindicated;
* Subjects who had already participated in an Org25969 trial;
* Subjects who had participated in another clinical trial (not pre-approved by NV Organon) within 30 days of entering into CT 19.4.310.
* Female subjects who are pregnant:
* Female subjects of childbearing potential not using any method of birth control: condom or using only hormonal contraception as birth control;
* Female subjects who were breast -feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2005-11-10 (Actual); Primary Completion 2006-05-22 (Actual); Study Completion 2006-08-29 (Actual)

PRIMARY OUTCOMES:
Time from start administration of Org 25969/neostigmine to recovery T4/T1 ratio to 0.9 | After surgery

SECONDARY OUTCOMES:
Time from start administration of Org 25969/neostigmine to recovery T4/T1 ratio to 0.7 and 0.8 | After surgery
Assessment of clinical signs of recovery (level of consciousness, 5 sec head lift, and general muscle weakness) | after surgery

REFERENCES:
- [Result] Flockton EA, Mastronardi P, Hunter JM, Gomar C, Mirakhur RK, Aguilera L, Giunta FG, Meistelman C, Prins ME. Reversal of rocuronium-induced neuromuscular block with sugammadex is faster than reversal of cisatracurium-induced block with neostigmine. Br J Anaesth. 2008 May;100(5):622-30. doi: 10.1093/bja/aen037. Epub 2008 Apr 2. PMID 18385265
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html